CLINICAL TRIAL: NCT06777329
Title: Standardization of the Dry Immersion Model Used as a Ground-based Model to Mimic Weightlessness. Part 3: a Comparison Study Between 10 Days of Dry Immersion vs. 10 Days of Head-down Bedrest on 20 Healthy Male Volunteers (VIVALDI 3)
Brief Title: A Comparison Study Between 10 Days of Dry Immersion Versus 10 Days of Head-down Bedrest on 20 Healthy Male Volunteers
Acronym: VIVALDI 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre National d'Etudes Spatiales (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 24-336; 2024-A02109-38 (Other: Agence Nationale de Sécurité du Médicament et des Produits de Santé (ANSM))
Record Dates: First submitted 2024-12-20; First posted 2025-01-15 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Weightlessness Simulation
Keywords: Comparison of 2 weightlessness simulation models
MeSH Terms: interventions — Head-Down Tilt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dry Immersion arm (Experimental): 10 days of dry immersion
  Interventions: Behavioral: 10 days of dry immersion
- Bed rest arm (Experimental): 10 days of head down bed rest
  Interventions: Behavioral: 10 days of Head Down Bed Rest

INTERVENTIONS:
Behavioral: 10 days of dry immersion — The volunteers in this arm will be immersed up to the neck for 10 days in a specially designed bath filled with tap water.
  Other Names: Dry Immersion (DI)
  Arms: Dry Immersion arm
Behavioral: 10 days of Head Down Bed Rest — The volunteers in this arm will spend 10 days in -6° head down bed rest.
  Other Names: Head Down Tilt (HDT)
  Arms: Bed rest arm

SUMMARY:
The space agencies are actively engaged in studying the physiological adaptation to space environment through studies on board the International Space Station (ISS) but also on the ground. Different methods are used to simulate weightlessness on Earth, including cellular models, animal models using hind-limb unloading, or on humans with unilateral lower limb suspension. However, two approaches, -6° head-down bed rest (HDBR) and dry immersion (DI) have provided possibilities for long-term exposures with findings closest to those seen with a weightless state. They produce changes in body composition (including body fluid redistribution), cardiovascular and skeletal muscle characteristics that resemble the effects of microgravity.

The common physiological denominator is the combination of a cephalad shift of body fluids and reduced physical activity. Being similar in their effects on the human body, these models, however, differ in their specifics and acting factors.

The Head-down Bedrest (HDBR) model has been widely used for this purpose and is considered one of the references for reproducing the physiological effects of weightlessness on Earth. During HDBR, subjects are lying down with an angle of -6° between the feet and head, on their side, their back or their front, but must keep one shoulder in contact with the mattress. All daily activities and tests are performed in this position.

One of the advantages of the HDBR model is that it has now been used in a great number of studies internationally, and its effects have long been described and compared with those of microgravity and spaceflight. Long-term bedrest is the gold-standard method for studying the effects of weightlessness and to test countermeasures.

Dry immersion involves immersing the subject in water covered with an elastic waterproof fabric. As a result, the immersed subject, who is freely suspended in the water mass, remains dry. Within a relatively short duration, the model can faithfully reproduce most physiological effects of actual microgravity, including centralization of body fluids, support unloading, and hypokinesia.

The objective of the present study is to compare the physiological adaptations to10 days of dry immersion versus 10 days of head-down bedrest in 20 healthy male subjects. A set of measurements will assess the changes in the cardiovascular, neuro-ophthalmological, hematological, metabolic, sensorimotor, immune, muscle and bone systems as a result of both models. The most likely outcome of this study will not be to show a clear superiority of one model over the other. Rather, we expect to show differences in kinetics and intensity of adaptations, that should vary from one system to another. This will help future researchers choose the best model depending on the system they are investigating and the rapidity or intensity of the effect they are exploring. The two models, instead of competing with one another, are probably complementary.

ELIGIBILITY:
* Healthy male volunteer (see below the description of medical tests and laboratory analysis performed at the selection visit),
* Age 20 to 40,
* No overweight nor excessive thinness with BMI (weight kg/ height m2) between 20 and 26,
* Height between 165cm and 180 cm,
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination): in particular, free from any chronic disease or any acute infectious disease or cardiovascular, neurological, ENT (especially orthostatic hypotension and vestibular disorders), orthopaedic or musculoskeletal disorders,
* Fitness level assessment: 35 ml/min./kg < VO2max < 55 ml/min./kg,
* Non active smokers,
* No alcohol, or drug addiction, and no medical treatment,
* Covered by a Health Insurance System,
* Having signed the informed consent,
* Free from any engagement during the study.

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, neurological or ENT (especially orthostatic hypotension and vestibular disorders), any chronic disease; any acute infectious disease. Particularly:
* Symptomatic orthostatic hypotension whatever the decrease in blood pressure, or asymptomatic postural hypotension defined by a decrease in SBP equal to or greater than 20 mmHg within 3 minutes when changing from the supine to the standing position,
* Cardiac rhythm disorders,
* Hypertension,
* Chronic back pains,
* Vertebral fracture, scoliosis or herniated disc,
* Glaucoma,
* Self-reported hearing problems,
* History of migraines,
* History of hiatus hernia or gastro-esophageal reflux,
* History of thyroid dysfunction, renal stones, diabetes,
* History of head trauma,
* History of genetic muscle and bone diseases of any kind,
* Past records of thrombophlebitis, family history of thrombosis or positive response in thrombosis screening procedure (anti thrombin III, S-protein, C-protein, factor V Leiden mutation and the mutation 20210 of the prothrombin gene),
* Signs of venous insufficiency, varicose veins, or telangiectasia
* Bone mineral density: T-score ≤ -1.5,
* Poor tolerance to blood sampling,
* Having given whole blood (more than 7ml/kg) in a period of 8 weeks or less before the start of the experiment, or having given whole blood more than 5 times in the past 12 months,
* Significant history of allergy, especially no dermatological allergy,
* History of food allergy,
* Significant anomaly detected in the biological analysis,
* Positive reaction to any of the following tests: HVA IgM (hepatitis A), HBs antigen (hepatitis B), anti-HVC antibodies (hepatitis C), anti-HIV1+2 antibodies,
* Vegetarian or vegan,
* Refusal to give permission to contact his general practitioner,
* Subject who, in the judgment of the investigator, is likely to be non-compliant during the study, or unable to cooperate because of a language problem or poor mental development,
* Subject already participating or in the exclusion period of a clinical research,
* Subject who has received more than 6000 Euros within 12 months for being a research subject,
* MRI contraindications:
* History or active claustrophobia,
* Osteosynthesis material, presence of metallic implants or any other contra-indication for MRI,
* Allergy to Gadolinium.
* Vulnerable persons according to law "Code de la Santé Publique" (L1121-5 to L1121-8) :
* Persons deprived of their liberty by an administrative or judicial decision,
* Persons under involuntary psychiatric care,
* Persons admitted in a health or social establishment for purposes other than research,
* Minors,
* Adults subject to legal protection (subject under guardianship or trusteeship) or unable to express their consent.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Changes in orthostatic tolerance | At baseline and first day of recovery
  Orthostatic tolerance (min) will be assessed during a progressive Lower Body Negative Pressure test (LBNP test)
Changes in peak aerobic power (VO2max test) | At baseline and the first day of recovery
  Exercise capacity (ml/kg/min) wil be assessed by graded cycling on sitting ergometer until exhaustion
Change in plasma volume | At baseline and 3 days after the end of the intervention
  Plasma volume (L) will be assessed by the carbon monoxide-rebreathing method
Change in plasma volume percentage | At baseline and at day 1, day 3, day 7 and at the end of the intervention periods
  The percentage change in plasma volume versus baseline (%) will be assessed by the Dill and Costill method
Change in fluid shift distribution towards the cardiac and cephalic region | At baseline, the first day to quantify the short term effect, the fifth day and the tenth day of interventions to quantify the long term effect of fluid shift
  The consequences of the fluid shift on the cardiac and cephalic area will be assessed by quantifying the carotid and femoral diameters (mm), as well as the carotid intima media thickness (mm) by ultrasound.
Change in body fluid compartments by bioelectrical impedance analysis | At baseline, during the ten days of intervention and until 3 days after the end of the intervention
  Extracellular, intracellular and total body water (L) will be estimated by bioimpedance
Change in calf and thigh circumferences | At baseline, during the intervention period and until 3 days after the intervention period
  Change in calf and thigh circumferences will be measured using a measuring tape (cm)
Change in fat and lean body mass measured by dual energy x-ray absorptiometry (DEXA) | At baseline, after 10 days of dry-immersion and 10 days of reovery
  Change in fat and lean body mass (g) measured by dual energy x-ray absorptiometry (DEXA)
Change in Resting Metabolic Rate (RMR) | At baseline, at day 3 and day 9 days of intervention periods
  RMR (kcal/24h) will be measured by indirect calorimetry technique
Change in nitrogen balance | At baseline, at day 3 and day 9 days of intervention periods
  Nitrogen balance is a measure of nitrogen input minus nitrogen output. Nitrogen intake (g) is calculated with a nutrition software. Total urinary nitrogen (g) in the 24-Hour urine collection estimates nitrogen output
Change in glucose tolerance (Oral Glucose Tolerance Test) | At baseline, at day 3 and day 9 days of intervention periods
  Glucose (mmol/L) levels will be measured at baseline (fasting) and 30, 60, 90, 120 and 180 minutes after drinking within 5 min a water solution containing 75 g of glucose
Change in serum bone formation marker (bone-specific Alkaline Phosphatase bAP) | At baseline and during the 10 days of interventions
  Change in bone-specific Alkaline Phosphatase (bAP, µg/L) will be assessed by chemiluminescence immunoassay
Change in serum bone resorption marker (C-terminal cross-linked telopeptide of type I collagen CTx) | At baseline and during the 10 days of interventions
  Change in C-terminal cross-linked telopeptide of type I collagen (CTx, pmol/L) will be assessed by chemiluminescence immunoassay will be assessed by enzyme-immmuno assay
Changes in bone density (by DEXA and High Resolution Peripheral Computed Tomography (HR-pQCT)) | At baseline and at day 10 of intervention periods
  Bone density (g/cm2) is measured at lumbar and hip level with DEXA and at tibia and radius level with HR-pQCT. Additionally tibia mechanical properties will be estimated by cortical ultrasound propagation velocity (m/s) via intraosseous ultrasonography.
Change in serum cartilage synthesis biomarkers | At baseline, during the intervention period and until 3 days after the intervention period
  Change in serum CP II and in human cartilage glycoprotein-39 (YKL-40) concentrations
Change in serum cartilage degradation biomarkers | At baseline, during the intervention period and until 3 days after the intervention period
  Change in serum Cartilage Oligomeric Matrix Protein (COMP) and fragments or propeptide of type II collagen (C2C, C1,2C, Coll-2-1) concentrations
Change in muscle strength | At baseline and after one day of recovery
  Muscle strength will be assessed from single leg isometric maximal voluntary contraction on the knee extensors & flexors, the plantarflexors and dorsiflexors. The Isometric Torque will be measured in Nm. The peak of the three maximal attempts will be recorded for strength measures
Changes in jump performance | At baseline and the first day of recovery
  Jump performance will be assessed on a platform and height of the jump will be evaluated
Change in contraction time | At baseline and at the end of the intervention periods
  Contraction time will be assessed during a measurement using the tensiomyography method in the following muscles: vastus lateralis, Gastrocnemius medialis and Biceps femoris of dominant leg.
Change in standing balance | At baseline and at day 1 and day 2 of recovery
  Standing balance (CoP velocity, mm/s) will be assessed by posturography eyes open and eyes closed on a platform covered with 12-cm thick medium density foam
Change in walking balance | At baseline and after 10 days of intervention and day 1 after the end of the intervention
  Functional mobility test (such as sit and walk, heel to toe steps with eyes closed and open, Triangle Completion Task) will assess walking balance.
Change in height | At baseline and at day 1, day 2 and day 3 of recovery
  Change in height (mm) measured in standing position
Change in mid cerebral artery (MCA) blow flow velocity | At baseline and one day after the intervention period
  Mid cerebral artery (MCA) blow flow velocity will be measured by transcranial Doppler
Change in circadian rhythms of blood pressure | At baseline and during the ten days of the intervention periods
  Continuous 24-h recording of systolic and diastolic blood pressure will be performed by a Non Invasive Blood Pressure system (SOMNOtouch™NIBP) designed for ambulatory continuous measurements
Change in mood | At baseline, at day 5 of the intervention period and 3 days after the end of the intervention
  Change in mood is assessed using the Profile of Mood States (POMS) questionnaire, by calculation of total mood disturbance (scale from -32 to 200, a higher score indicates more severe mood disturbance)
Change in affective states | At baseline, at day 5 of the intervention period and 3 days after the end of the intervention
  Positive and Negative Affect Schedule (PANAS) questionnaire will be used to assess the intensity of positive (range from 10 to 50, with higher scores representing higher levels of positive affect) and negative (range from 10 to 50, with lower scores representing lower levels of negative affects) affective states. PANAS self-report questionnaire consists of two 10-item scales to measure both positive and negative affects.
Change in sleep quality | Daily from baseline to 10 days after the end of the intervention
  Pittsburgh Sleep Dairy (PghSD) will be used to assess sleep perceived quality. The PghSD is an instrument with separate components to be completed at bedtime and waketime. The following parameters are registered or assessed:
  Bedtime, waketime, sleep latency, wake after sleep onset, total sleep time, mode of awakening and ratings of sleep quality, mood, and alertness on wakening, as well as daytime information on naps, exercise, meals and caffeine, tobacco and medications use.
Change in psychological state: mental health | At baseline, at day 5 of the intervention period and 4 days after the end of the intervention
  ical well-being and capture distress
  GHQ-28 gives an overall total score and 4 scores for 4 subscales:
  Somatic symptoms, Anxiety/insomnia, Social dysfunction, Severe depression. Higher scores indicate higher levels of distress
Change in coping strategies | At day 5 of the intervention and 2 days after the end of the intervention
  Brief Cope Questionnaire is designed to measure effective and ineffective ways to cope with a stressful life event, and will be used to assess coping strategies. The Brief Cope is a shortened form (28 items) of the Carver and Scheier COPE inventory.
  There are 14 coping strategies. These strategies can be then gathered in two main categories : approach coping and avoidance coping.
Measurement of changes in subjective sleepiness | At baseline, at day 4 and 8 of the intervention period and 3 days after the end of the intervention
  Changes in subjective level of sleepiness will be measured using the Karolinska sleepiness scale (KSS) two times per day, with a scale from 1 to 10 (higher scores reprensent higher sleepiness).
Change in circadian variations of heart rate | At baseline, at day 1, day 4, day 7 of intervention, and at first day of recovery
  Difference between day-time and night-time heart rate (bpm) will be calculated
Change in daily body movements | Continuously from baseline until 5 days after the intervention period
  Accelerometry-derived daily physical activity counts will be quantified using actigraph GT3X+
Dynamics of body fluids during the 4 first hours of exposure | The 4 first hours of Dry Immersion / Bed Rest
  Changes from pre to 240 min of exposure for plasma volume percentage versus baseline (%) assessed by the Dill and Costill method
Lower limb vascular properties | At baseline, at day 10 of intervention periods, and day 3 of recovery
  Change in tibial intracortical blood flow velocity (mm/s), induced by physiological maneuvers (velocity of intracortical blood flow at medial tibia level and its responses to vascular occlusion will be assessed via Ultrasound Vector Flow Mapping)
Myofiber atrophy | At baseline and at day 8 of intervention
  Biopsy sampling from m. vastus lateralis will be performed. Myofiber CSA related to fiber type (µm2) will be measured by morphometric analysis.
Post-occlusive reactive hyperemia at great toe and thumb level | At baseline and 4 days after the end of the intervention
  Blood flow (AU) will be assessed via Laser Doppler flowmetry. Post-occlusive reactive hyperemia index will be calculated.
Quantitative sensory testing at the dorsum of the foot (vibration detection threshold) | At baseline, at day 7 of intervention periods, and day 2 of recovery
  Vibration detection threshold (s) will be measured using graded tuning fork
Whole-body MRI | At baseline, at day 9 of intervention periods
  Change in MRI-measured whole-body Lean mass (kg) and Fat mass (kg) will be estimated
Vestibular health evaluation | At baseline and the first day of recovery
  Battery of tests routinely performed on astronauts will be used. Sit-to-stand time (s) will be quantified.
Blood cytokines evolution | At baseline, at day 3 & 10 of intervention periods, and day +10 of recovery
  To characterize immune functions, the following blood cytokines (pg/ml) will be assessed: TPO, G-CSF, IL-1β, IL-1Ra, IL-4, IL-6, IL-8, IL-10, IFNy, TNF
Salivary cortisol evolution | At baseline, at day 1, 3 & 10 of intervention periods, and day +4 & +10 of recovery
  To characterize stress level, morning and evening salivary cortisol (ng/ml) will be assessed
Change in optic nerve sheath diameter (ONSD) considered as an indirect marker for intracranial pressure (ICP) estimation | From baseline to 1 day after the end of the intervention
  The optic nerve sheath diameter (ONSD) variations will be measured by echography
Change in intraocular pressure (IOP) | From baseline to 1 day after the end of the intervention
  IOP measured by applanation
Change in visual acuity | At baseline and 2 days after the intervention period
  Far and near visual acuity are tested uncorrected, or if applicable with own correction with digital acuity system
Change in visual field | At baseline and 2 days after the intervention period
  Visual field measured by standard automated perimetry
Change in the anatomical characteristics of the eye (optical biometry) | At baseline and 2 days after the intervention period
  Optical biometry measured by partial coherence interferometry
Change in the central corneal thickness | At baseline and 2 days after the intervention period
  Central corneal thickness on a single point on the cornea measured by Ultrasonic pachymetry
Change in the retina by non-mydriatic fundus retinography | At baseline and 2 days after the intervention period
  Non-mydriatic fundus retinography allows a fundus photography to be taken and thus a color image of the papilla, retinal vessels and macula
Change in the cornea topography | At baseline and 2 days after the intervention period
  Cornea topography measured by corneal topography equipment (like Pentacam). The elevation topography according to Scheimpflug principle allows the mapping of the anterior and posterior surface of the cornea.
Change in cerebral structures and in venous circulation of the brain by MRI | At baseline and at day 9 of intervention
  Visualization of cerebral structures and intracranial venous system will be performed by MRI coupled with injection of gadolinium
Change in thrombotic and fibrinolytic processes | At baseline, during the intervention and 2 days after the intervention period
  Thrombotic and fibrinolytic processes will be assessed by thromboelastometry (TEM, coagulation analyzer from Matel Medizintechnik, Graz, Austria), providing a kinetic analysis of the clot formation process and of clot dissolution by the fibrinolytic system. Clotting time (min) wil be measured.
Change in energy requirements | At baseline and at day 2 of the intervention period
  Change in energy requirements using the doubly labelled water
Change in skin microcirculation | At baseline and 3 days after the intervention period
  Indirect evaluation of cardiovascular and neurovascular change by performing deep inspiration. Blood flow (AU) at great toe will be assessed via Laser Doppler flowmetry. Inspiratory gasp vascular response (%) will be calculated.
Change in cardiovascular deconditioning and orthostatic tolerance (stand test) | At baseline and 2 days after the intervention period
  This test continuously measures heart rate (bpm) via a Finapres device while subjects sit for 5 minutes, then stand for 5 minutes and then sit again for 5 minutes
Change in stress and mental load | From baseline to 10 days after the end of the intervention
  This test assesses the effects of dry immersion and bed rest on cognitive tasks involving various executive functions (e.g., attention, memory, decision-making) by assessing both physiological (via the SOMNO HD system) and behavioral parameters (e.g., emotions, cognitive load) using the D2 test of attention. Pourcentage of errors (%) will be measured as a qualitative aspect of performance.

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Antoine CUSTAUD, MD, PhD, Study Director — University Hospital, Angers
Locations (1):
- Medes-Institut de Médecine et de Physiologie Spatiale, Toulouse, France, France